CLINICAL TRIAL: NCT05987007
Title: Sleep Interventions and Neurocognitive Outcomes in Amnestic Mild Cognitive Impairment
Brief Title: Sleep Interventions and Neurocognitive Outcomes
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: Columbia University (Other)
Responsible Party: Principal Investigator, Hyun "Monica" Kim, Assistant Professor of Clinical Psychology, New York State Psychiatric Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 8443
Record Dates: First submitted 2023-05-22; First posted 2023-08-14 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Sleep Disturbance; Amnestic Mild Cognitive Impairment
Keywords: Alzheimer's Disease; Slow-Wave Activity; Older Adults; Amnestic Mild Cognitive Impairment; Cognitive Behavioral Therapy for Insomnia
MeSH Terms: conditions — Parasomnias; Alzheimer Disease | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Cognitive Behavioral Therapy for Insomnia (Active Comparator): Participants assigned to the CBTI treatment group will receive 8 weeks of weekly telehealth sessions with a masters-level therapist. Each session is approximately 50 minutes in duration.
  Interventions: Behavioral: Cognitive behavioral therapy for insomnia
- Acoustic Slow-Wave Activity Enhancement (Active Comparator): Participants assigned to the SWAE group will be instructed to use the Dreem2 headband at least four nights out of seven nights of the week.
  Interventions: Device: Acoustic slow-wave activity enhancement

INTERVENTIONS:
Device: Acoustic slow-wave activity enhancement — The acoustic enhancement of slow-wave activity will be conducted using the Dreem2 headband. This device utilizes five dry-EEG electrodes (O1, O2, FpZ, F7, and F8), a 3D accelerometer, and a pulse oximeter to detect slow-wave activity and generates acoustic stimulation of slow-waves to augment slow-wave sleep.
  Arms: Acoustic Slow-Wave Activity Enhancement
Behavioral: Cognitive behavioral therapy for insomnia — Cognitive behavioral therapy for insomnia (CBTI) is a well-established first-line or complimentary treatment for insomnia which consists of cognitive and behavioral modifications, including addressing maladaptive sleep-related behaviors, controlling sleep environment, and limiting time spent in bed.
  Arms: Cognitive Behavioral Therapy for Insomnia

SUMMARY:
This protocol focuses on the effect of sleep interventions on improving sleep and building cognitive/brain resilience in older adults with amnestic mild cognitive impairment and sleep disturbance. Two sleep interventions, cognitive behavioral therapy for insomnia (CBTI) and acoustic slow-wave activity enhancement (SWAE), will be utilized in a pilot randomized clinical trial in which participants are randomized to different treatment groups (CBTI or SWAE). Participants will be assessed over a 6-month period in order to examine the impact of sleep treatments on neuropsychological outcomes and cognitively mediated everyday functioning.

DETAILED DESCRIPTION:
This study has the goal of understanding the effect of sleep interventions on improving sleep and building cognitive/brain resilience in older adults. To implement this, the investigators will conduct a pilot randomized clinical trial in which fifty older adults (with amnestic mild cognitive impairment and sleep disturbance) will be assigned to different treatment groups to test the effects of cognitive behavioral therapy for insomnia (CBTI) and acoustic slow-wave activity enhancement (SWAE) over the course of 6 months. CBTI is a psychotherapy intervention designed to address maladaptive cognitive and behavioral patterns associated with sleep and bedtime. SWAE is administered through a non-invasive headband that detects and amplifies endogenous slow-wave activity using playing acoustic stimulation ("pink noise"). Group differences will be compared on the changes in cognitive performance and plasma biomarkers of Alzheimer's disease (phosphorylated tau). The investigators will also explore potential mechanisms behind the relationship between sleep and cognition/biomarkers by investigating a range of objectively measured sleep metrics (e.g., sleep architecture, sleep duration, arousals) along with APOE genotype and depressive symptoms.

ELIGIBILITY:
Inclusion Criteria:

1. English speaking participants, ages 60-85 years
2. Telephone MMSE (T-MMSE) score of 22 or greater at screening assessment; T-MMSE <18 during post-treatment visit or 6-month follow-up will be discontinued from participation of the study.
3. Individuals with aMCI, as determined by the Wechsler Memory Scale-Revised Logical Memory Delayed Recall (LM) and Quick Dementia Rating Scale (QDRS)
4. Presence of subject memory complains not exclusionary. Presence of subjective memory complaints without objective signs of impairment (T-MMSE, QDRS, LM) would not be considered as the presence of late MCI or dementia, therefore are not exclusionary.
5. Participants with regular and consistent use of sleep medications (sedatives/hypnotic use of >3 times per week) will be excluded. Participants who take sleep medications 3 or less times per week will be asked to discontinue medications prior to the study baseline visit. All discontinuation/tapering procedures will require PI's direct consultation with participants' prescribing or primary care physicians, which will be documented to ensure participants' safety.
6. Presence of sleep disturbance, as determined by score of 8 or greater on the Insomnia Severity Index administered at baseline (without sleep medications).
7. Participants must have capacity to provide informed consent.
8. Have access to stable internet connection.
9. A family member or other individual who is in contact with the subject and consents to serve as informant during the study; this can be a telephone informant in the case of subjects who do not have a live-in informant

Exclusion Criteria:

1. Diagnosis of stroke or excessive risk of CVD
2. Neurologic disease including movement disorders, MS, epilepsy, and TBI (with greater than 15 min loc)
3. Untreated diabetes
4. Active treatment of cancer
5. Telephone MMSE score below 22 (Newkirk et al., 2004) and Logical Memory above 11 for subjects with 16 or more years of education, 9 for subjects with 8-15 years of education, and 6 for subjects with 0-7 years of education
6. Presence of sleep disorders other than insomnia (moderate-severe sleep apnea, REM-behavior disorder, restless legs syndrome, circadian rhythm disorder). Mild sleep apnea will not be exclusionary.
7. Current DSM-5 Axis I psychiatric diagnosis of schizophrenia, schizoaffective disorder, substance/alcohol use disorder, or bipolar disorder
8. Use of antidepressants with known large anticholinergic properties will be excluded. These include: amitriptyline, amoxapine, clomipramine, desipramine, doxepine, imipramine, isocarboxazide, lithium, maprotiline, mirtazapine, nortriptyline, tranylcypromine trimipramine, and phenelzine. Other medications are allowed during the study and are not exclusionary.
9. Participants taking medications with benzodiazepines properties will be excluded. These include: diazepam, quazepam, estazolam, alprazolam, clorazepate, clorazepate, oxazepam, alprazolam, chlordiazepoxide, lorazepam, flurazepam, triazolam, temazepam, and midazolam.
10. Participants with moderate to severe depression (Geriatric Depression Scale>8) will be excluded from the study and will be encouraged to seek treatment for their symptoms. Participants with moderate depression (GDS 5-8) will be encouraged to return for screening after receiving treatment and seeing improvement in their symptoms.
11. Participants who are unable to provide an informant.

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
No Practice Effect (NPE) battery | Baseline, Week 9, Week 24
  The total composite score, as well as factor scores (Cognitive Control and Executive Functions, Episodic Memory Consolidation, Verbal Working Memory) will be examined.
Everyday Cognition (ECog) | Baseline, Week 9, Week 24
  Total score and subdomains (Everyday Planning, Everyday Organization, Everyday Divided Attention, Everyday Language, Everyday Visuospatial Abilities, Everyday Memory Subdomain scores) will be examined.
Conners Continuous Performance Test (CPT-3) | Baseline, Week 9, Week 24
  Measure of sustained attention and vigilance

SECONDARY OUTCOMES:
Insomnia Severity Index | Baseline, Week 9, Week 24
  Well-established measure of insomnia symptoms. Scores range from 0-28, and higher scores represent more severe insomnia symptoms.
N3 sleep stage ("slow-wave sleep") | Baseline, Week 9, Week 24
  N3 sleep duration will be calculated using Dreem Headband, a sleep assessment device that produces objective sleep measures.
SubjectiveTotal Sleep Time | Baseline, Week 9, Week 24
  Self-reported sleep duration will be asked as part of the sleep diaries.
Objective Total Sleep Time | Baseline, Week 9, Week 24
  Objective sleep duration will be measured via sleep monitoring device (Dreem Headband 2)
Subjective Wake After Sleep Onset | Baseline, Week 9, Week 24
  Self-reported sleep duration will be asked as part of the sleep diaries.
Objective Wake After Sleep Onset | Baseline, Week 9, Week 24
  Objective sleep duration will be measured via sleep monitoring device (Dreem Headband 2)

CONTACTS AND LOCATIONS:
Overall Officials: Hyun Kim, PhD, Principal Investigator — Columbia University/ New York State Psychiatric Institute
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
All subject data will be de-identified. Clinical trial data with accompanying metadata, and bio-samples (if relevant) will be housed at GAAIN, a publicly available data repository funded and maintained by the Alzheimer's Association and will comply with all standard practices for data management. As defined within PAR-21-359 for early-stage clinical trials, all study data, including post-randomization trial data, raw and processed primary data, and remaining bio-samples (if relevant), will be made available to the scientific community at the time of publication of the primary results or within 9 months of database lock, whichever comes first. We will provide the necessary documentation, metadata, and supporting information to ensure proper understanding and utilization of the shared data.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: At the time of publication of the primary results or within 9 months of database lock, whichever comes first.
Access Criteria: Requests are made and detailed using a 2-page request form with the following sections:
  Significance; Data Requested; Methodologies; Statistical Plan; Alignment with study goals.
  Data request review criterion:
  The review criteria will include the significance of the request; use of appropriate methodologies; absence of conflict with other on-going data analysis by our group or outside investigators already conducting similar studies; and alignment with the basic goal of the grant (cognitive enhancement in aMCI and understanding its mechanisms).
  We will provide progress reports to the NIH on data sharing activities, including the number of data access requests received, approved, and denied, as well as updates on the utilization and impact of the shared data.